CLINICAL TRIAL: NCT04403971
Title: Effect of 0.12% Chlorhexidine Oral Care for the Prevention of Non-ventilator Hospital-acquired Pneumonia Among Hospitalized Patients
Brief Title: 0.12% Chlorhexidine Oral Care for the Prevention of Non-ventilator Hospital-acquired Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chen, Yen-Chin, Vice Head Nurse and Clinical Assistant Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: A-ER-108-309
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Hospital-acquired Pneumonia
Keywords: 0.12% chlorhexidine; Oral rinse; Hospital-acquired pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.12% chlorhexidine (Experimental): Participants will be randomized to Chlorhexidine solution group, applied twice a day by care givers.
  Interventions: Drug: 0.12% Chlorhexidine Oral Liquid Product
- Listerine (Sham Comparator): Participants will be randomized to Listerine solution group, applied twice a day by care givers.
  Interventions: Drug: Listerine Oral Liquid Product
- Normal saline (Placebo Comparator): Participants will be randomized to Normal saline group, applied twice a day by care givers.
  Interventions: Other: Normal Saline Product

INTERVENTIONS:
Drug: 0.12% Chlorhexidine Oral Liquid Product — The intervention group 1 received 10ml 0.12% chlorhexidine solution for oral rinse twice a day.
  Arms: 0.12% chlorhexidine
Drug: Listerine Oral Liquid Product — The intervention group 2 received 10ml Listerine solution for oral rinse twice a day.
  Arms: Listerine
Other: Normal Saline Product — The control group received 10ml normal saline for oral rinse twice a day.
  Arms: Normal saline

SUMMARY:
Chlorhexidine is a effective strategy in reducing ventilator associated pneumonia. However, it is unclear if prophylactic 0.12% chlorhexidine oral rinse can reduce the risk of non-ventilator hospital-acquired pneumonia among hospitalized patients.

DETAILED DESCRIPTION:
Participants will be classified into three groups, applied twice a day by care givers. Oral colonization will be tested in the baseline, day-3, day-7, and at the discharge. Quantitation of colonization of the oral cavity by oral rinses and respiratory pathogens were measured.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients > 20 years old without ventilator

Exclusion Criteria:

* known hypersensitivity to or intolerance of Chlorhexidine or Listerine

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
oral bacterial colonization status | 1 year

SECONDARY OUTCOMES:
The rate of non-ventilator associated pneumonia | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Yen-Chin Chen, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sangmuang P, Lucksiri A, Katip W. Factors Associated with Mortality in Immunocompetent Patients with Hospital-acquired Pneumonia. J Glob Infect Dis. 2019 Jan-Mar;11(1):13-18. doi: 10.4103/jgid.jgid_33_18. PMID 30814830
- [Background] Giuliano KK, Baker D, Quinn B. The epidemiology of nonventilator hospital-acquired pneumonia in the United States. Am J Infect Control. 2018 Mar;46(3):322-327. doi: 10.1016/j.ajic.2017.09.005. Epub 2017 Oct 16. PMID 29050905
- [Background] Quinn B, Baker DL, Cohen S, Stewart JL, Lima CA, Parise C. Basic nursing care to prevent nonventilator hospital-acquired pneumonia. J Nurs Scholarsh. 2014 Jan;46(1):11-9. doi: 10.1111/jnu.12050. Epub 2013 Sep 30. PMID 24119253
- [Background] Chou CC, Shen CF, Chen SJ, Chen HM, Wang YC, Chang WS, Chang YT, Chen WY, Huang CY, Kuo CC, Li MC, Lin JF, Lin SP, Ting SW, Weng TC, Wu PS, Wu UI, Lin PC, Lee SS, Chen YS, Liu YC, Chuang YC, Yu CJ, Huang LM, Lin MC; Infectious Diseases Society of Taiwan;; Taiwan Society of Pulmonary and Critical Care Medicine,; Medical Foundation in Memory of Dr. Deh-Lin Cheng;; Foundation of Professor Wei-Chuan Hsieh for Infectious Diseases Research and Education;; CY Lee's Research Foundation for Pediatric Infectious Diseases and Vaccines,; 4th Guidelines Recommendations for Evidence-based Antimicrobial agents use in Taiwan (GREAT) working group. Recommendations and guidelines for the treatment of pneumonia in Taiwan. J Microbiol Immunol Infect. 2019 Feb;52(1):172-199. doi: 10.1016/j.jmii.2018.11.004. Epub 2018 Dec 6. PMID 30612923
- [Background] Zhang J, Ab Malik N, McGrath C, Lam O. The effect of antiseptic oral sprays on dental plaque and gingival inflammation: A systematic review and meta-analysis. Int J Dent Hyg. 2019 Feb;17(1):16-26. doi: 10.1111/idh.12331. Epub 2018 Feb 6. PMID 29405627